CLINICAL TRIAL: NCT05486806
Title: Longitudinal Tracking of Patients Diagnosed With Neurodegenerative Movement Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Vikram Khurana, MD PhD, Chief, Division of Movement Disorders, Brigham and Women's Hospital
Other Study IDs: 2022P001295
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Neurodegenerative Diseases; sca3; MSA - Multiple System Atrophy; Ataxia; Synucleinopathies
MeSH Terms: conditions — Neurodegenerative Diseases; Muscular Disorders, Atrophic; Shy-Drager Syndrome; Ataxia; Synucleinopathies | interventions — N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participants: all participants in this study must have a diagnosis of a neurodegenerative movement disorder
  Interventions: Drug: 18F-PBR06; Radiation: 18F-PBR06

INTERVENTIONS:
Drug: 18F-PBR06 — TSPO-PET (translocatior protein, positron emission tomography) scan
Radiation: 18F-PBR06 — TSPO-PET (translocatior protein, positron emission tomography) scan

SUMMARY:
The purpose of this protocol is to create an active natural history cohort of patients with degenerative movement disorders, tracked in a clinical setting with clinical rating scales and neuroimaging. The overarching rationale is that neurodegenerative diseases may be heterogeneous, complex disorders. A new way of performing clinical trials in these patients may be in order and this protocol aims to build a longitudinally tracked clinical trial-ready cohort of patients. The purpose of this protocol is to establish an active natural history cohort of patients with neurodegenerative movement disorders who are deeply phenotyped and "clinical trial ready" across Mass General Brigham.

After a thorough clinical diagnostic evaluation (this may include clinically indicated testing, for example MRI, FDG-PET, MIBG scan, polysomnography, genetic testing, autonomic function tests, inflammatory tests, skin biopsy) the investigators aim to achieve this through:

1. Longitudinal tracking of clinical progression through use of clinical scales including at the present time: UMSARS, BARS, MoCA and UPSIT, PROM, MDS-NMS, UPDRS, and SARA
2. Longitudinal tracking of disease progression through use of neuroimaging including at the present time: TSPO-PET and 3D MRI (see section 1.3)

This is a pilot study designed to track patients with neurodegenerative movement disorders across Mass General Brigham through MRI and PET imaging modalities and clinical measures. Figure 5 represents the study design in detail. In short, subjects will be asked to visit Mass General Brigham every 6-9 months over the course of 18 months for imaging and clinical evaluation.

DETAILED DESCRIPTION:
After a thorough clinical diagnostic evaluation (this may include clinically indicated testing, for example MRI, FDG-PET, MIBG scan, polysomnography, genetic testing, autonomic function tests, inflammatory tests, skin biopsy) the investigators aim to achieve this through:

1. Longitudinal tracking of clinical progression through use of clinical scales including at the present time: UMSARS, BARS, MoCA and UPSIT, PROM, MDS-NMS, UPDRS, and SARA
2. Longitudinal tracking of disease progression through use of neuroimaging including at the present time: TSPO-PET and 3D MRI (see section 1.3)

This is a pilot study designed to track patients with neurodegenerative movement disorders across Mass General Brigham through MRI and PET imaging modalities and clinical measures. Figure 5 represents the study design in detail. In short, subjects will be asked to visit Mass General Brigham every 6-9 months over the course of 18 months for imaging and clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of neurodegenerative movement disorder by consensus criteria including: MSA, ataxias, synuclein duplication, atypical parkinsonism
2. Male and female subjects aged 18 and up

Exclusion Criteria:

1. Individuals with a known alternate neurologic disorder including: idiopathic PD, DLB, PSP, ALS, Alzheimer's, prion disease, frontotemporal dementia, seizure disorder, stroke, or brain tumor
2. Individuals with a previous head injury (with 15 minutes or greater loss of consciousness within the past 20 years)
3. Individuals with substance abuse, or substance abuse disorder
4. Brain MRI indicative of a significant abnormality (i.e. prior hemorrhage or infarct greater than 1 cm3, 3 or more lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space- occupying lesion).
5. Individuals with bipolar disease and schizophrenia
6. Concurrent medical conditions that contraindicate study procedures
7. Women who are pregnant, nursing, or seeking to become pregnant
8. Individuals with claustrophobia
9. Non-MRI compatible implanted devices
10. Corticosteroid treatment in the past four weeks
11. Low affinity binders to TSPO
12. Significant cognitive impairment (MoCA score ≤ 23) or poor understanding of study design

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: individuals with a clinical diagnosis of neurodegenerative movement disorder by consensus criteria (MSA, ataxias, synuclein duplication, atypical parkinsonism, etc)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
association between change in PET and clinical measures | 18 months
  For the longitudinal evaluation, the investigators will estimate the association between the change in the PET and the change in the clinical and morphometric outcome measures using a mixed model with both the baseline PET uptake and the rate of change in PET uptake as predictors. This approach will allow the investigators to estimate both how between and within subject changes in PET impact the outcomes of interest. The investigators will use a p<0.05, corrected for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Khurana, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No